CLINICAL TRIAL: NCT03723941
Title: Mitotane With or Without Cisplatin and Etoposide After Surgery in Treating Participants With Stage I-III Adrenocortical Cancer With High Risk of Recurrence
Brief Title: Adjuvant Chemotherapy vs. Observation/Mitotane After Primary Surgical Resection of Localized Adrenocortical CarcInoma
Acronym: ACACIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alfredo Berruti, Head of Oncology Unit, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACACIA; ADIUVO-2 (Other: MD Anderson)
Record Dates: First submitted 2018-10-09; First posted 2018-10-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; Adjuvant Chemotherapy
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Cisplatin; Etoposide; Chemotherapy, Adjuvant; Observation; Mitotane

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, stratified, nation-based multi-center, phase III trial for patients with ACC and Ki67≥10% after resection with curative intent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - adjuvant therapy (Experimental): adjuvant therapy with four cycles of cisplatin plus etoposide +/- mitotane according to investigator's preference versus
  Interventions: Drug: Cisplatin plus Etoposide; Other: Observation or Mitotane
- B - observation or mitotane alone (Other): observation or mitotane alone according to the investigator's preference
  Interventions: Other: Observation or Mitotane

INTERVENTIONS:
Drug: Cisplatin plus Etoposide — Etoposide 100 mg/m2 will be administered IV on days 1, 2, 3 diluted in 500 mL of isotonic NaCl or 5% dextrose.
  Cisplatin, 80 mg/m2 will be administered IV on day 1, diluted in 500 mL of isotonic NaCl.
  Other Names: Adjuvant Chemotherapy
  Arms: A - adjuvant therapy
Other: Observation or Mitotane — Observation or mitotane alone according to the investigator's preference

SUMMARY:
Adrenocortical carcinoma (ACC) is a rare endocrine malignancy. Despite complete resection of early-stage disease recurrence rates in ACC are very high (60%.70%). Patients with Ki67 ≥ 10% are considered at high risk for ACC recurrence, whereas patients with Ki67<10% are considered to have low/intermediate risk for recurrence. No study are ongoing on adjuvant systemic therapy in ACC patients that are at high risk of relapse. These patients represent 70-80% of all ACC radically operated. In this setting mitotane is widely prescribed. The efficacy of mitotane is known to be dependent on the attainment of serum drug levels in the so called therapeutic range that is above 14 mg/l. However, ACC patients with high relapse risk may develop disease recurrence before mitotane serum levels attain the target concentration. Chemotherapy with cisplatin containing regimen was shown to be efficacious in the management of ACC in few phase II trials. Based on the background, there is a strong rationale of administering chemotherapy in radically operated ACC patients with high risk of relapse defined as follows: stage I-III ACC (according to the ENSAT classification) with either microscopically complete resection (R0), microscopically positive margins (R1), or undetermined margins (RX) and Ki67≥10% (for a further definition of this condition, see the study population paragraph). In clinical practice, adjuvant mitotane alone or cisplatin-based chemotherapy or the combination of both are used worldwide in patients at high risk of relapse, but there is no prospective validation of these treatments. The investigators will test the efficacy of the combination of cisplatin plus etoposide (plus/minus mitotane according to the investigator preference) in comparison with the actual best routine practice consisting of mitotane or no therapy (according to the personal belief of clinical investigator). This study is parto of the international trial registry ADIUVO-2 coordinated by MD Anderson Center of Huston (Texas).

DETAILED DESCRIPTION:
Adrenocortical carcinoma (ACC) is a rare endocrine malignancy with an annual rate of 0.5.2 cases per million population. Despite complete resection of early-stage disease recurrence rates in ACC are very high (60%.70%). Patients with Ki67 ≥ 10% are considered at high risk for ACC recurrence, whereas patients with Ki67<10% are considered to have low/intermediate risk for recurrence. Due to rarity of the disease no data from randomized clinical trials are available on the efficacy of any adjuvant therapies. Mitotane has been widely used in the adjuvant setting in ACC on the basis of the findings of a retrospective multicenter report in which relapse free survival (RFS) was significantly prolonged in patients treated with adjuvant mitotane compared with two control groups who were not given mitotane. The retrospective design of this study resulted in controversy about the benefit of adjuvant mitotane and led to a prospective clinical trial to compare mitotane to placebo as adjuvant therapy in low-risk/intermediate-risk ACC patients who have low Ki67 expression (<10%; ADIUVO study, ClinicalTrials.gov Identifier: NCT00777244).

No study are ongoing on adjuvant systemic therapy in ACC patients that are at high risk of relapse. These patients represent 70-80% of all ACC radically operated. In this setting mitotane is widely prescribed. The efficacy of mitotane is known to be dependent on the attainment of serum drug levels in the so called therapeutic range that is above 14 mg/l. These mitotane levels should be maintained over time. The results of a recent retrospective analysis on the impact of serum mitotane levels on prognosis in 122 ACC patients, who were radically resected, showed that the 63 patients who reached and maintained the target mitotane concentrations during follow-up had a significantly lower rate of recurrence than the 59 patients who failed to keep mitotane levels as high. However, the attainment of therapeutic range of mitotane usually require 2-3 months whatever is the schedule adopted. ACC patients with high relapse risk may develop disease recurrence before mitotane serum levels attain the target concentration.

Chemotherapy with cisplatin containing regimen was shown to be efficacious in the management of ACC in few phase II trials.

The results of the only phase III trial conducted up to now, the FIRM-ACT study, found that mitotane combined with cisplatin-based chemotherapy was superior to mitotane combined with streptozocin in terms of progression free survival and overall survival in patients with advanced/metastatic ACC. The cytotoxic activity of chemotherapy is rapid and this is the rationale of administering a cisplatin containing regimen in adjuvant setting of ACC patients with high risk of disease relapse.

Adjuvant mitotane treatment improved RFS and overall survival (OS) in a retrospective study, and adjuvant mitotane is undergoing prospective evaluation in low-risk/intermediate-risk ACC patients (Ki67<10%; ADIUVO study). However, Mitotane alone could be not adequate as adjuvant therapy in highly proliferating ACC since the drug efficacy is strictly dependent on the attainment of circulating concentration levels >14 mg/l that is usually achieved after 2-3 months of therapy. In this lead time disease recurrence may occur.

Based on the background, there is a strong rationale of administering chemotherapy in radically operated ACC patients with high risk of relapse defined as follows: stage I-III ACC (according to the ENSAT classification) with either microscopically complete resection (R0), microscopically positive margins (R1), or undetermined margins (RX) and Ki67≥10% (for a further definition of this condition, see the study population paragraph). In clinical practice, adjuvant mitotane alone or cisplatin-based chemotherapy or the combination of both are used worldwide in patients at high risk of relapse, but there is no prospective validation of these treatments.

In this multicenter prospective randomized clinical study, that will test the efficacy of the combination of cisplatin plus etoposide (plus/minus mitotane according to the investigator preference) in comparison with the actual best routine practice consisting of mitotane or no therapy (according to the personal belief of clinical investigator). This proposed randomized prospective study is needed to assess the efficacy and safety of chemotherapy with a cisplatin regimen in high-risk ACC patients after initial surgical resection. There are no studies ongoing testing any adjuvant therapies in radically operated ACC with high risk of relapse and death.

STUDY DESIGN AND DURATION

The study is designed as a prospective, randomized, open-label, stratified, nation-based multi-center, phase III trial for patients with ACC and Ki67≥10% after resection with curative intent.

Patients will be stratified on the basis of the European Network for the Study of Adrenal Tumors (ENSAT) stage (I/II vs. III) and whether the clinical investigator decide to administer mitotane or not.

The evaluation of ACC recurrence with imaging techniques (TC scan or MR) will be performed every 4 months for the first 2 years and then every 6 months till the 4th year.

In this study, the planned patient enrollment time is two years and the follow-up time is one year.

An international large scale prospective randomized clinical trial with a similar design of the present study is currently being submitted to national and international calls for funds. If this trial will be funded and will start, the present trial will converge to the international one, and the funds obtained by AIFA wil be employed to manage the italian part.

STUDY POPULATION

The patients that will be enrolled in this study will have newly diagnosed and radically operated ACC at high risk of disease recurrence defined as follows:

* stage I-III ACC (according to the ENSAT classification) AND
* Ki67≥10%

SAMPLE SIZE

The sample size calculation is performed on the basis of the following assumption. The median RFS for the mitotane group with Ki67≥10% is estimated to be 20 months. It is assume that Cisplatin + Etoposide therapy can reduce the risk of disease recurrence or death assuming a median RFS of 34 months for arm A, which translates into a hazard ratio (Cisplatin + Etoposide [+/- mitotane] vs. observation [+/- mitotane] of 0.59, and a drop-off rate of 5% in each arm. Therefore, a total sample size of 198 patients (rounded to 200, 100 in each arm) is needed to achieve a power of 80% to detect an improvement in median RFS of 14-months (from 20 months to 34), with a one-sided significance level of 0.05 and an interim analysis when 1/3 of events will be recorded. The study duration is expected to be about 3 years: 2-years for recruitment and 1-year of minimum follow-up. The Clinical Epidemiology Unit - Clinical Trial Center of the Città della Salute e della University Hospital in Turin, will provide a web based procedure for randomization and a dedicated database for eCRF (www.epiclin.it).

METHODS

Etoposide 100 mg/m2 will be administered IV on days 1, 2, 3 diluted in 500 mL of isotonic NaCl or 5% dextrose over 60 minutes.

Cisplatin, 80 mg/m2 will be administered IV on day 1, diluted in 500 mL of isotonic NaCl, over 60 minutes. Before cisplatin, 1000 ml isotonic NaCl with addition of 20 mmol potassium is given during 2 h. Cisplatin infusion is administered over 60 minutes. Cisplatin administration is followed by 1000 ml isotonic NaCl with addition of 5 mmol Magnesium and 20 mmol potassium during 1 hour. 500 mL mannitol IV can also be administered at a concentration of 150 mg/mL during 1 hour according to the inestigator routine clinical practice. Injections of small doses of diuretics (e.g. furosemide 10-20 mg) should be given IV to ensure diuresis and avoid retention of fluids.

Cisplatin and etoposide regimen will be administered every 21 days for 4 cycles.

Treatment should start within 7 days from randomization. If the clinical investigator decide to prescribe mitotane (alone or in combination with chemotherapy according to the randomization treatment arm), the drug will be administered orally to reach a plasma level of 14.20 mg/L (or the maximum tolerated dose if unable to reach therapeutic levels). The mitotane dosage scheme is the responsibility of the local investigator, but an initial dose of 3.6 g daily is usually prescribed to reach therapeutic plasma mitotane levels (14.20 mg/L). Dosage will be further adjusted according to blood concentrations and clinical assessment.

Analysis of serum mitotane levels will be performed monthly by a reputable clinical laboratory chosen by each center to reflect clinical practice patterns. All patients on mitotane will receive concomitant glucocorticoid replacement therapy with the option of using plasma adrenocorticotropic hormone levels to guide steroid replacement.

Mitotane will be administered to the two study arms until ACC relapse, intolerable toxicity, or for a total period of 2 years.

RANDOMIZATION

The randomization procedure will be performed online and implemented with the electronic case report form at the web-site www.epiclin.cpo.it.

The procedure will be stratified on the following factors:

Mitotane use Disease stage (I/II vs. III) Ki67 percentage (10%.20% vs. >20%)

SCHEDULED VISITS AND PROCEDURES

The baseline evaluation (1 week before randomization) includes:

History and physical examination Concomitant medications Surgical and pathological reports Complete blood count Serum biochemistry profile, lipid profile Endocrine assessment: serum cortisol, testosterone (in women), 17-hydroxyprogesterone, dehydroepiandrosterone sulfate, aldosterone, estradiol (in men and postmenopausal women), adrenocorticotropic hormone (ACTH), plasma renin activity, free T4, and TSH Pregnancy test in women of childbearing potential every 3 months or if there is suspicion for pregnancy EKG CT with contrast (or MRI) of the chest/abdomen/pelvis performed no more than 4 weeks before randomization Written informed consent After the completion of baseline procedures, the patient will be randomized.

The subsequent visits will be as follows:

1. Arm A (cisplatin+etoposide +/- mitotane): in the first 12 weeks after randomization, clinical visits every 3 weeks (±3 days) will include:

   Physical examination Report of side effects and concomitant medications CBC Serum chemistry profile Endocrine assessment Serum mitotane evaluation (if applicable)
2. Arm B (mitotane or observation): in the first 12 weeks after randomization, every 4 weeks, clinical visits will include:

Physical examination Report of concomitant medications If the patient is receiving mitotane the following data will be requested Report of side effects CBC Serum chemistry profile Endocrine assessment Serum mitotane measurement At 16 weeks (in both study arms), and every 16 weeks until ACC recurrence cross-sectional imaging studies (MRI or CT with contrast medium) of the chest/abdomen/pelvis will be performed. Further imaging can be ordered if deemed necessary by the local investigator (CT or MRI of the brain or bone assessment).

After the first 12 weeks (in both study arms) until ACC recurrence: Every 12 weeks, the clinical visit will include:

Physical examination Report of concomitant medications and side effects CBC Serum chemistry profile Endocrine assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ACC (Weiss score of ≥ 3); all tumor specimens can be reviewed a posteriori by a reference pathologis
* High risk of relapse within 60 days of surgical resection of primary tumor with curative intent with either microscopically complete resection (R0, microscopically positive margins (R1), or undetermined margins (RX, based on surgical or pathological reports without unequivocal evidence of metastasis in the perioperative imaging).
* Ki67≥10% (to be determined by an experienced pathologist in each participating center and preferably via quantitative imaging analysis).
* Have perioperative imaging (CT with contrast or MRI of the chest/abdomen/pelvis) demonstrating no unequivocal evidence of disease within 4 weeks before randomization. Patients with indeterminate non-specific nodules (<1 cm for soft tissue lesions and <1.5 cm in the short dimension for lymph nodes) will be permitted to participate in this study.
* Be 18 years old or older.
* Have a negative pregnancy test no more than 7 days before starting treatment
* Adequate contraception
* Have an Eastern Cooperative Oncology Group performance status 0.2
* Have an adequate bone marrow reserve (neutrophils >1,000/mm3 and/or platelets >80,000/mm3)
* Have an adequate organ function (including renal, liver and cardiac function)
* Be able to comply with the protocol procedures and provide written informed consent.

Exclusion Criteria:

* The time between primary surgery and randomization is >60 days
* They have undergone repeated surgery for recurrence of disease
* They have a history of recent or active prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, breast ductal carcinoma in situ, or other treated malignancies where there has been no evidence of disease for at least 2 years
* They have renal insufficiency (estimated glomerular filtration rate [GFR] <50 mL/min/1.73 m2) or significant liver insufficiency (serum bilirubin>2 times the upper normal range and/or serum alanine aminotransferase [ALT] or aspartate aminotransferase [AST]>3 times the upper normal range). GFRs will be calculated according to the validated formula (MDRD)
* They are pregnant or breast feeding
* They have congestive heart failure (ejection fraction<45%). In patients with a history of cardiac disease, a baseline two-dimensional echocardiogram is needed to document ejection fraction. In patients without prior cardiac disease, a baseline electrocardiogram (EKG) is sufficient if there is no evidence of acute ischemic changes or prior evidence of myocardial infarction. If EKG results are abnormal (ischemic changes, significant arrhythmia, or suggestion of prior myocardial infarction), a two-dimensional echocardiogram will be obtained to assess ejection fraction
* They have preexisting grade 2 peripheral neuropathy
* They underwent previous or current treatment with mitotane or other antineoplastic drugs for ACC
* They underwent previous radiotherapy for ACC
* They have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration or that, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the recurrence-free survival (RFS) status in patientis treated with adiuvant chemotherapy with or without mitotane (arm A) versus no treatment or adjuvant mitotane (arm B). | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Evaluation of recurrence-free survival (RFS). Recurrence will be objectively assessed every 16 weeks by imaging the chest/abdomen/pelvis by either computed tomography (CT; with slice thickness of 5 mm or less) or magnetic resonance imaging (MRI). Suspected lesions will be accurately measured in at least one dimension (the longest diameter in the plane of measurement will be recorded). Soft tissue lesions must have a minimum size of 10 mm, and suspected malignant lymph nodes must be more than 15 mm (short axis) to be considered pathological.

SECONDARY OUTCOMES:
Assessment of overal survival | From date of randomization until the date of death from any cause, assessed up to 36 months
  defined as the time interval between the date of randomization and the date of death from any cause.
Assessment of toxicity and adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Toxicity and adverse events will be graded according to the NCI-CTCAE (version 4.03).
Assessment of the predictive role of Ki67 expression for chemotherapy efficacy | Ki67 expression evaluated at the screening phase
  Histological evaluation of KI67 expression on basal tumor tissue sections and correlation to chemotherapy efficacy
Assessment of the predictive role of histopathologic characteristics (Weiss-score) for chemotherapy efficacy | Weiss score identified at the screening phase
  Weiss score will be identified on basal tumor tissue resection based on the original Weiss criteria for malignancy (Am J Surg Pathol 1984;8:163), and will be correlated to chemotherapy efficacy. The Weiss scoring system is based on the recognition at light microscopy of nine morphological parameters: three of them are related to tumor structure, namely presence of eosinophilic ("dark") cytoplasm in more than 75% of tumor cells, of a "patternless" diffuse architecture, and of necrosis; three others are related to cytological features, namely presence of nuclear atypia, of mitotic index above 5 per 50 high-power fields, and of atypical mitoses; the remaining three are related to invasive tumor properties, including sinusoidal, venous, and capsular invasion. A diagnosis of malignancy is achieved if at least three parameters are identified out of 9 (scale from 0 to 9).

OTHER OUTCOMES:
BioBank | Baseline
  Available tissue specimens (formalin-fixed paraffin-embedded or frozen tissues) plus one sample of serum, plasma and urine, will be collected before randomization for each patient enrolled in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kebebew E, Reiff E, Duh QY, Clark OH, McMillan A. Extent of disease at presentation and outcome for adrenocortical carcinoma: have we made progress? World J Surg. 2006 May;30(5):872-8. doi: 10.1007/s00268-005-0329-x. PMID 16680602
- [Result] Grubbs EG, Callender GG, Xing Y, Perrier ND, Evans DB, Phan AT, Lee JE. Recurrence of adrenal cortical carcinoma following resection: surgery alone can achieve results equal to surgery plus mitotane. Ann Surg Oncol. 2010 Jan;17(1):263-70. doi: 10.1245/s10434-009-0716-x. Epub 2009 Oct 23. PMID 19851811
- [Result] Beuschlein F, Weigel J, Saeger W, Kroiss M, Wild V, Daffara F, Libe R, Ardito A, Al Ghuzlan A, Quinkler M, Osswald A, Ronchi CL, de Krijger R, Feelders RA, Waldmann J, Willenberg HS, Deutschbein T, Stell A, Reincke M, Papotti M, Baudin E, Tissier F, Haak HR, Loli P, Terzolo M, Allolio B, Muller HH, Fassnacht M. Major prognostic role of Ki67 in localized adrenocortical carcinoma after complete resection. J Clin Endocrinol Metab. 2015 Mar;100(3):841-9. doi: 10.1210/jc.2014-3182. Epub 2015 Jan 5. PMID 25559399
- [Result] Berruti A, Baudin E, Gelderblom H, Haak HR, Porpiglia F, Fassnacht M, Pentheroudakis G; ESMO Guidelines Working Group. Adrenal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii131-8. doi: 10.1093/annonc/mds231. No abstract available. PMID 22997446
- [Result] Terzolo M, Angeli A, Fassnacht M, Daffara F, Tauchmanova L, Conton PA, Rossetto R, Buci L, Sperone P, Grossrubatscher E, Reimondo G, Bollito E, Papotti M, Saeger W, Hahner S, Koschker AC, Arvat E, Ambrosi B, Loli P, Lombardi G, Mannelli M, Bruzzi P, Mantero F, Allolio B, Dogliotti L, Berruti A. Adjuvant mitotane treatment for adrenocortical carcinoma. N Engl J Med. 2007 Jun 7;356(23):2372-80. doi: 10.1056/NEJMoa063360. PMID 17554118
- [Result] Terzolo M, Fassnacht M, Ciccone G, Allolio B, Berruti A. Adjuvant mitotane for adrenocortical cancer--working through uncertainty. J Clin Endocrinol Metab. 2009 Jun;94(6):1879-80. doi: 10.1210/jc.2009-0120. No abstract available. PMID 19494162
- [Result] Hermsen IG, Fassnacht M, Terzolo M, Houterman S, den Hartigh J, Leboulleux S, Daffara F, Berruti A, Chadarevian R, Schlumberger M, Allolio B, Haak HR, Baudin E. Plasma concentrations of o,p'DDD, o,p'DDA, and o,p'DDE as predictors of tumor response to mitotane in adrenocortical carcinoma: results of a retrospective ENS@T multicenter study. J Clin Endocrinol Metab. 2011 Jun;96(6):1844-51. doi: 10.1210/jc.2010-2676. Epub 2011 Apr 6. PMID 21470991
- [Result] Terzolo M, Baudin AE, Ardito A, Kroiss M, Leboulleux S, Daffara F, Perotti P, Feelders RA, deVries JH, Zaggia B, De Francia S, Volante M, Haak HR, Allolio B, Al Ghuzlan A, Fassnacht M, Berruti A. Mitotane levels predict the outcome of patients with adrenocortical carcinoma treated adjuvantly following radical resection. Eur J Endocrinol. 2013 Jul 29;169(3):263-70. doi: 10.1530/EJE-13-0242. Print 2013 Sep. PMID 23704714
- [Result] Senkus E, Kyriakides S, Penault-Llorca F, Poortmans P, Thompson A, Zackrisson S, Cardoso F; ESMO Guidelines Working Group. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi7-23. doi: 10.1093/annonc/mdt284. Epub 2013 Aug 22. No abstract available. PMID 23970019
- [Result] Berruti A, Terzolo M, Pia A, Angeli A, Dogliotti L. Mitotane associated with etoposide, doxorubicin, and cisplatin in the treatment of advanced adrenocortical carcinoma. Italian Group for the Study of Adrenal Cancer. Cancer. 1998 Nov 15;83(10):2194-200. PMID 9827725
- [Result] Bonacci R, Gigliotti A, Baudin E, Wion-Barbot N, Emy P, Bonnay M, Cailleux AF, Nakib I, Schlumberger M; Reseau Comete. Cytotoxic therapy with etoposide and cisplatin in advanced adrenocortical carcinoma. Br J Cancer. 1998 Aug;78(4):546-9. doi: 10.1038/bjc.1998.530. PMID 9716042
- [Result] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- [Result] Tsuchiya R, Suzuki K, Ichinose Y, Watanabe Y, Yasumitsu T, Ishizuka N, Kato H. Phase II trial of postoperative adjuvant cisplatin and etoposide in patients with completely resected stage I-IIIa small cell lung cancer: the Japan Clinical Oncology Lung Cancer Study Group Trial (JCOG9101). J Thorac Cardiovasc Surg. 2005 May;129(5):977-83. doi: 10.1016/j.jtcvs.2004.05.030. PMID 15867769
- [Result] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Result] Oberg K. Chemotherapy and biotherapy in the treatment of neuroendocrine tumours. Ann Oncol. 2001;12 Suppl 2:S111-4. doi: 10.1093/annonc/12.suppl_2.s111. PMID 11762335
- [Result] Brix D, Allolio B, Fenske W, Agha A, Dralle H, Jurowich C, Langer P, Mussack T, Nies C, Riedmiller H, Spahn M, Weismann D, Hahner S, Fassnacht M; German Adrenocortical Carcinoma Registry Group. Laparoscopic versus open adrenalectomy for adrenocortical carcinoma: surgical and oncologic outcome in 152 patients. Eur Urol. 2010 Oct;58(4):609-15. doi: 10.1016/j.eururo.2010.06.024. Epub 2010 Jun 22. PMID 20580485
- [Result] Habra MA, Ejaz S, Feng L, Das P, Deniz F, Grubbs EG, Phan A, Waguespack SG, Ayala-Ramirez M, Jimenez C, Perrier ND, Lee JE, Vassilopoulou-Sellin R. A retrospective cohort analysis of the efficacy of adjuvant radiotherapy after primary surgical resection in patients with adrenocortical carcinoma. J Clin Endocrinol Metab. 2013 Jan;98(1):192-7. doi: 10.1210/jc.2012-2367. Epub 2012 Nov 12. PMID 23150683